CLINICAL TRIAL: NCT01171872
Title: Gene Expression in Inflammatory Bowel Disease
Status: Enrolling by invitation | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: NA_00038329; U01DK062431 (NIH); R24DK099803 (NIH); P01AI125181 (NIH)
Record Dates: First submitted 2010-07-28; First posted 2010-07-29 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Inflammatory Bowel Disease
Keywords: Inflammatory Bowel Disease; Inflammatory Bowel Disease (IBD); Crohn's Disease; Ulcerative Colitis; Indeterminate Colitis; IBD; CD; UC; IC
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood, serum, tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Unaffected: Individuals who do not have IBD
- Affected: Individuals who have IBD

SUMMARY:
Inflammatory bowel disease (IBD), including Crohn's disease (CD) and ulcerative colitis (UC), is a idiopathic, chronic and frequently disabling inflammatory disorder of the intestines characterized by a dysregulated mucosal immune response that affect more than a million Americans. This protocol is aimed at obtaining tissue samples to test for expression of genes associated with IBD and to better understand the pathogenesis of IBD with the study of genetics, proteomics, physiologic processes and microbiomes (microbiology).

DETAILED DESCRIPTION:
Progress has been made in recent years in understanding the pathological mechanisms of IBD, particularly in the search of IBD susceptibility genes. However, due to the extreme complexity of the diseases, there is still a long way ahead in elucidating detailed molecular mechanisms of IBD pathogenesis and identifying more effective therapeutic targets. Therefore, it is the goal of this research study to discover genetic, microbial, gene expression and serological factors involved in the pathogenesis of IBD which may pave the way for the identification of more effective therapeutic targets.

The specific aims for these objectives are as follows:

AIM 1: Identify proteins that are changed in expression and post-translational modification in the intestinal mucosa of patients with active UC or CD compared to i) uninvolved intestinal mucosa from the same patients, ii) normal intestinal mucosa in control subjects, and iii) infectious/Inflammatory colitis (C. difficile colitis).

AIM 2: Identify changes in the expression of intestinal membrane transporters for Na absorption and Cl secretion, including NHE3, in the intestinal mucosa of patients with active UC or CD compared to i) uninvolved intestinal mucosa from the same patients, ii) normal intestinal mucosa in control subjects, and and iii) infectious/Inflammatory colitis (C. difficile colitis). The targeted screening will also include several intestinal epithelial brush border-associated PDZ-containing proteins that have been recently shown to regulate trafficking and activity of membrane transporters.

AIM 3: Enteroid Sub-study - To compare the physiologic regulation of Na absorption, Cl secretion, protein secretion and other intestinal physiologic processes in IBD cases, other infectious colitis cases and healthy controls as these processes are often altered with disease activities. The processes will be studied through the development of self-propagating culture models called organoids or enteroids. The culture models are developed from biopsy specimens taken from the upper small intestine, including duodenum and jejunum , lower small intestine (ileum) and proximal and distal colon and used to grow organoids/enteroids. These are mini-intestines that have the entire crypt villus axes which grow in culture and can be kept alive indefinitely in culture.

AIM 4: Mechanism of Intestinal Inflammation Sub-study - To understand the mechanisms involved in the recurrence of inflammation following ileal resection surgery for Crohn's disease (CD). Reasons for recurrence are currently unknown but are believed to be caused by an interaction of genetic, immune and microbial features. Information gained from this study will be used to build a predictive model to identify those patients at greater risk of rapid recurrence, and will aid physicians in tailoring follow-up treatments.

AIM 5: UC Demarcation Sub-study - To gain further understanding of the mechanisms involved in the susceptibility to and flare of inflammation in UC patients. Blood, stool, urine, saliva, lavage and tissue samples from UC patients will be used to help study the genetic, microbial, metabolic, and immune factors involved in the remission and flare of disease. Information gained from this study will also be used to build a predictive model of which patients are at greater risk of disease flare, and which are less likely to do so, allowing physicians to tailor follow-up treatments accordingly.

ELIGIBILITY:
Inclusion Criteria:

* All persons, regardless of IBD affection status, greater than 7 years of age undergoing upper or lower endoscopy or bowel resection

Exclusion Criteria:

* Persons with bleeding tendencies
* Persons on anti-coagulation therapy or who will be place on anti-coagulation therapy following the planned endoscopy procedures

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals who are to undergo upper or lower gastrointestinal endoscopies or a surgical resection as part of their normal medical care and deemed necessary by their physicians.
  Patients are primarily recruited at the Johns Hopkins inpatient and outpatient units. However, individuals can contact us by phone, mail or email after hearing about our study.
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 1999-11 (Actual); Primary Completion 2032-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Gene Expression in IBD | Single visit, approximately 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Florin Selaru, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States